CLINICAL TRIAL: NCT07399119
Title: The Immediate Effect of Adding the Wim Hoff Breathing Method With Aerobic Training on Aerobic Performance and Hemodynamic Response in Smoking Adults
Brief Title: The Study Examined the Acute Effects of Wim Hof on Aerobic Training and Cardiodynamics.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Takey Ahmed, Khaled Takey Ahmed - Associateprofessor, Cairo University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-H-0237-HSC-R-0763 - BAU.
Record Dates: First submitted 2026-01-15; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Abnormality; Pulmonary; Exercise Training
Keywords: wim hoff; aerobic
MeSH Terms: interventions — Jogging

STUDY DESIGN:
Intervention Model Description: stop watch - blood pressure monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): Researchers took the first measurement at t=0 minutes after 5 minutes of their arrival to allow them to rest. The measurements included heart rate and SpO2 using an oximeter (Medical Rossmax) and blood pressure using a sphygmomanometer. Then they were asked to perform a 12-minute walk/jog with speed controlled by them and incline = 1. At 4 and 8 minutes, the speed was reduced to 2.0 on the treadmill, and vitals were taken again. At t= 12 minutes we stopped the treadmill, recorded the distance covered, and proceeded to measure the heart rate. SpO2, blood pressure, and VO2max were calculated using the Cooper's test formula (Alvero-Cruz et al., 2017). Participants were asked to rest for 4 minutes, and then another measurement of the vital signs (heart rate, SpO2, and blood pressure) was taken before they were dismissed.
  Interventions: Other: aerobic exercise where it included walking/ jogging with a controlled speed by the participant
- wim hof breathing exercises (Experimental): applying breathing interventions
  Interventions: Other: aerobic exercise where it included walking/ jogging with a controlled speed by the participant; Other: Wim Hof Breathing Method

INTERVENTIONS:
Other: aerobic exercise where it included walking/ jogging with a controlled speed by the participant — participants were asked to listen attentively to the given instruction using noise cancelling headphones for the given instructions. For 11 minutes, an audio for Wim Hof breathing method that is as follow.
  * Take a strong inhalation through the nose.
  * Let out a relaxed exhalation through the mouth.
  * Repeat for 30 breaths.
  * On the 30th breath, exhale and hold your breath for 30 seconds in the first round then 1 minute in the 2nd round and 1 and a half minutes for the 3rd round.
  * Take a deep breath in after the previous hold then hold it in for 15 seconds in the 3 rounds.
  * Let your breathing return to normal. These steps were repeated for 3 rounds. And participants were allowed to let go of their held breath and hold it again if they couldn't keep holding it for the asked time in the audio
Other: Wim Hof Breathing Method — participants were asked to listen attentively to the given instruction using noise cancelling headphones for the given instructions. For 11 minutes, an audio for Wim Hof breathing method that is as follow.
  * Take a strong inhalation through the nose.
  * Let out a relaxed exhalation through the mouth.
  * Repeat for 30 breaths.
  * On the 30th breath, exhale and hold your breath for 30 seconds in the first round then 1 minute in the 2nd round and 1 and a half minutes for the 3rd round.
  * Take a deep breath in after the previous hold then hold it in for 15 seconds in the 3 rounds.
  * Let your breathing return to normal. These steps were repeated for 3 rounds. And participants were allowed to let go of their held breath and hold it again if they couldn't keep holding it for the asked time in the audio
  Arms: wim hof breathing exercises

SUMMARY:
Researchers will split the sixty healthy smokers in half. Thirty people will serve as a control group and will be asked to walk or jog at a controlled pace for twelve minutes as part of an aerobic exercise program. Separately, 30 people participated in an aerobic exercise session that lasted 12 minutes and involved walking or running at a pace that the participants themselves controlled. WHBM will be done both prior to and subsequent to physical activity. To determine how WHBM affects the experimental group's pre- and post-WHBM heart rates, SpO2, blood pressure, and VO2 max, this study will be conducted.

DETAILED DESCRIPTION:
The study will be a randomized single blinded control trial, sixty healthy smokers will be divided into two groups. a control group of 30 participants will performing a 12-minute aerobic exercise where it included walking/ jogging with a controlled speed by the participant. Another experimental group of 30 participants also, performing a 12-minute aerobic exercise where it included walking/ jogging with a controlled speed by the participant. WHBM will be performed before and after exercises. It will be done to assess the effect of WHBM on heart rate, SpO2, blood pressure and VO2 max that will be monitored before and after WHBM in the experimental group. In addition, Performance will be assessed by observing the difference in distance covered before and after doing the WHBM. Heart rate and SpO2 will be measured using a finger pulse oximeter (Medical Rossmax). Blood pressure will be measured using a sphygmomanometer and VO2 max will be measured using the cooper's test formula in kilometers: "VO2 max = (22.351 x distance in Km) - 11.288"

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* Age range between 18 and 25 years.
* Adults who are healthy

Exclusion Criteria:

If they had:

* Any systemic disorders.
* Musculoskeletal, neuromuscular, or chronic respiratory conditions.
* Females were menstruating

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
HEART RATE | 12 weeks
  The number of heartbeats in a minute
Vo2 max | 12 weeks
  oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: rami L abbass, professor, Study Director — BAU
Locations (1):
- BAU, Beirut, Tariq EL Jedida, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
measured data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 months

REFERENCES:
- See also: doi — https://doi.org/10.1371/journal.pone.0225749